CLINICAL TRIAL: NCT01489566
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multi-Center Phase III Clinical Trial to Evaluate the Safety and Efficacy of Injectable Tyroserleutide to Treat Hepatocellular Carcinoma
Brief Title: Study of Tyroserleutide for Injection in Hepatocellular Carcinoma (HCC) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Collaborators: Fudan University (Other); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYS-CN-1.1PUMP III
Record Dates: First submitted 2011-12-01; First posted 2011-12-09 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Hepatocellular,Carcinoma
Keywords: Hepatocellular,Carcinoma,recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — H-Tyr-Ser-Leu-OH; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tyroserleutide for injection (Active Comparator): the Tyroserleutide for injection at the dosage of 6mg/d
  Interventions: Drug: Tyroserleutide for injection ,chemotherapy(mitomycin, and Fluorouracil )
- the placebo (Placebo Comparator)
  Interventions: Drug: the placebo ,chemotherapy(mitomycin, and Fluorouracil )

INTERVENTIONS:
Drug: Tyroserleutide for injection ,chemotherapy(mitomycin, and Fluorouracil ) — mitomycin(10mg)+Fluorouracil(1.0g),through the chemoradiative pump,every cycle,5-30 minites; Tyroserleutide for injection(30mg) ,through the micro infusion pump,every cycle,3-5 days
  Arms: Tyroserleutide for injection
Drug: the placebo ,chemotherapy(mitomycin, and Fluorouracil ) — mitomycin(10mg)+Fluorouracil(1.0g),through the chemoradiative pump,every cycle,5-30 minites; the placebo(30mg) ,through the micro infusion pump,every cycle,3-5 days
  Arms: the placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi-center Clinical Trial. Patients with no tumor lesions one month after resection of hepatocellular carcinoma will be randomized in a 1:1 ratio to 1 of the 2 treatment groups：6mg/d Tyroserleutide (injection), or placebo.

The objective is to evaluate the effect of Injectable Tyroserleutide on the recurrence-free survival,overall survival,quality of life,and the safety and tolerability of subjects after the resection of hepatocellular carcinoma

DETAILED DESCRIPTION:
* Subjects will return to the hospital 25±5 days after the resection of hepatocellular carcinoma following the baseline examination. Baseline imaging data will be sent to the lead study site imaging center for review and verification. The investigator will determine whether the subject satisfies all inclusion/exclusion criteria. If all requirements are satisfied, then randomization will occur 25±5 days after surgery
* The day of randomization will be defined as Day 0. Randomized subjects will return to the hospital and begin cycle 1 on the day of randomization (Day 0). The Investigator will administer chemotherapy according to the subject's condition. On the next day, experimental drug therapy will begin, and the relevant laboratory tests will be performed within 3 days after the end the study drug infusion.
* Cycles will occur every four weeks for the first 6 cycles (i.e. cycles 2, 3, 4, 5, and 6 will begin on days 28 ± 3, 56 ± 3, 84 ± 3, 112 ± 3, and 140 ± 3, respectively). The second 6 cycles will occur every eight weeks (i.e. cycles 7, 8, 9, 10, and 11, will begin on days 196 ± 3, 252 ± 3, 308 ± 3, 364 ± 3, and 420 ± 3, respectively).
* the participant will receive medical inspection so as to observe and ensure drug safety.
* A CT scan will be performed for each participant to exclude the recurrence or metastasis of tumor and assess the effects of treatment once before the initiation of each new cycle.

ELIGIBILITY:
Perioperative Period Inclusion Criteria

1. Signed informed consent;
2. Aged ≥ 18 years and ≤ 75 years old, male or female；
3. Subject underwent a complete resection of hepatocellular carcinoma (confirmed by pathology);
4. The tumor characteristics must meet one of the following:

   * Tumor thrombosis in the portal vein branches is detected by either;

     * Preoperative imaging, or;
     * Intraoperative visual observation.
   * Tumor thrombosis in the portal vein branches was not detected; and

     * A single tumor with a maximum diameter ≥8cm confirmed by preoperative imaging, and histological evidence of micro vascular tumor thrombosis; or
     * Preoperative imaging confirmed that there are 2 or more tumor lesions

Perioperative Period Exclusion Criteria

1. Concomitant malignant primary tumor(s) in other systems is/are present;
2. Tumor thrombosis in the main branch of portal vein or in hepatic vein is detected by preoperative imaging or observed during the surgery;
3. The subject received any previous systemic anti-HCC therapy prior to the resection surgery (except the resection surgery), such as liver transplantation, intervention, ablation, radiotherapy, chemotherapy, molecular targeted therapy or other anti-HCC therapy;
4. The subject took other study/investigational drugs 7 days prior to the resection surgery;
5. The subject has central nervous system disease, mental illness, unstable angina, congestive heart failure, severe arrhythmia or other severe uncontrolled diseases;
6. The subject has history of study drug or similar drug allergy

Baseline (Post-SurgeryDay 25 ± 5) Inclusion Criteria

1. Baseline (post-resection) liver CT (normal CT + contrast enhanced CT) and chest CT scan show no tumor lesions;
2. Child-Pugh score of class A at baseline

Baseline (Post-SurgeryDay 25 ± 5) Exclusion Criteria

1. Body surface area is < 1.47 m2 or > 1.92 m2;
2. Concomitant malignant primary tumor(s) in other systems is/are present;
3. The subject took other study/investigational drugs within 4 weeks prior to randomization;
4. The baseline examination indicates that infection, bleeding, bile leakage, or other postoperative complications are present;
5. The baseline examination suggests the presence of tumor metastasis;
6. The subject has central nervous system disease, mental illness, unstable angina, congestive heart failure, severe arrhythmia or other severe uncontrolled diseases;
7. The subject has history of investigational drug or similar drug allergy;
8. The subject is pregnant, lactating, or urine pregnancy test result is positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
RFS(Recurrence Free Survival) | 0-2years
  The time from randomization to recurrence, metastasis or death due to any reason

SECONDARY OUTCOMES:
OS （Overall Survival） | 0-2years
  The time from randomization to death due to any reason
QOL score | 0-2years
  Quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Tang ZhaoYou, Academician, Study Chair — Shanghai Zhongshan Hospital; Wu Meng Chao, Academician, Study Chair — Second Milliary Medical University,Eastern Hepatobiliary Surgery Hosipital; Fan Jia, professor, Study Director — Shanghai Zhongshan Hospital; Yang Jia Mei, professor, Study Director — Second Milliary Medical University,Eastern Hepatobiliary Surgery Hosipital; Sun Hui Chuan, professor, Principal Investigator — Shanghai Zhongshan Hospital; Yan Yi Qun, professor, Principal Investigator — Second Milliary Medical University,Eastern Hepatobiliary Surgery Hosipital; Zheng Shu Sen, Academician, Principal Investigator — The First Affiliated Hospital of College of Medicine, Zhejiang Universtiy; Wu Yu Lian, professor, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine; Dong Jia Hong, professor, Principal Investigator — Chinese PLA General Hospital; Sang Xin Ting, professor, Principal Investigator — Peking Union Medical College Hospital; Chen Min Shan, professor, Principal Investigator — Sun Yat-sen University; Guo Rong Ping, professor, Principal Investigator — Sun Yat-sen University; Zheng Qi Chang, professor, Principal Investigator — Tongji Medical College,Huazhong University of Science and Technology Wuhan Union Hospital; Xia Xiao Qin, professor, Principal Investigator — Hubei Cancer Hospital; Liu Jing Feng, professor, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Chen Yan Ling, professor, Principal Investigator — Fujian Medical University Union Hospital; Ying Min Gang, professor, Principal Investigator — Fujian Cancer Hospital; Shi Xue Tao, professor, Principal Investigator — Shandong Cancer Hospital and Institute; Liu Jun, professor, Principal Investigator — Shandong Provincial Hospital; Liu Ji Yong, professor, Principal Investigator — Shandong Provincial Hospital; Wu Jin Shu, professor, Principal Investigator — Hunan Provincial People's Hospital; Wang Zhi Ming, professor, Principal Investigator — Xiangya Hospital of Central South University; Yang Xun, professor, Principal Investigator — Sichuan Provincial People's Hospital; Yan Lv Nan, professor, Principal Investigator — West China Hospital,Sichuan Universtiy; Bie Ping, professor, Principal Investigator — Southwest Hospital, China; Ma Kuan Sheng, professor, Principal Investigator — Southwest Hospital, China; Liu Qing Guang, professor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Han Ying, professor, Principal Investigator — Xijing Hospital; Wang Xue Hao, professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Ding Yi Tao, professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Hao Xi Shan, Academician, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Liu Lian Xin, professor, Principal Investigator — Center of First Affiliated Hospital of Harbin Medical University; Li Wei, professor, Principal Investigator — The First Affiliated Hospital of Jilin University; Wang Guang Yi, professor, Principal Investigator — The First Affiliated Hospital of Jilin University; Jiang Bo, professor, Principal Investigator — Hunan Provincial People's Hospital; Du Qin, professor, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China